CLINICAL TRIAL: NCT00000318
Title: Buprenorphine Maintenance Dose Schedule and Treatment Setting: Pilot
Brief Title: Buprenorphine Maintenance Dose Schedule and Treatment Setting - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Yale University (Other)
Responsible Party: Richard S. Schottenfeld, MD, Yale University School of Medicine
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-09803-1; R01-09803-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-12

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: opioid dependence
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Maintenance treatment with daily medication
  Interventions: Drug: Buprenorphine
- 2 (Experimental): Maintenance treatment with thrice-weekly medication
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — 1. Experimental Maintenance treatment with daily medication
  2. Experimental Maintenance treatment with thrice-weekly medication

SUMMARY:
The purpose of this study is to assess optimal dosage of buprenorphine on a thrice weekly schedule in a pilot clinical trial.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 1994-12; Primary Completion 2004-03 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Opioid and cocaine use | 26 weeks
Social and psychological functioning | 26 weeks
AIDS risk behavior | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schottenfeld, M.D., Principal Investigator — Yale University
Locations (1):
- APT Residential Services Division, New Haven, Connecticut, United States